CLINICAL TRIAL: NCT05784090
Title: Livelli di Melatonina e Dei Suoi Precursori/Metaboliti in Differenti Fluidi Biologici: vi è Correlazione?
Brief Title: Correlation Between Melatonin Levels in Different Biological Fluids
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 21C821
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Neurodegenerative Diseases
MeSH Terms: conditions — Neurodegenerative Diseases | interventions — Blood Specimen Collection; Spinal Puncture

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, saliva and cerebrospinal fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- AD: Alzheimer's Disease
  Interventions: Other: blood and saliva sample and lumbar puncture diagnostic for specific neurological diseases
- NON AD: Non Alzheimer's Disease
  Interventions: Other: blood and saliva sample and lumbar puncture diagnostic for specific neurological diseases
- CT: Controls
  Interventions: Other: blood and saliva sample and lumbar puncture diagnostic for specific neurological diseases

INTERVENTIONS:
Other: blood and saliva sample and lumbar puncture diagnostic for specific neurological diseases — Saliva was collected using Salivettes (Sarsted, Newton, NC, USA) in dim light. CSF was obtained in the morning after overnight fasting by lumbar puncture at the L3/L4 or L4/L5 interspace.
  Blood samples were drawn in fasting conditions. Plasma was separated by centrifugation.

SUMMARY:
The goal of this observational study is to evaluate and to correlate melatonin levels in plasma, saliva and cerebrospinal fluid (CSF) samples of patients undergoing lumbar puncture diagnostic for specific neurological diseases.

ELIGIBILITY:
Inclusion Criteria:

* Neurodegenerative disease

Exclusion Criteria:

* Age < 18 years
* Pregnancy
* Coagulations disorders
* Anticoagulant therapy

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Neurodegenerative disorders
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2018-10-23 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Melatonin levels in saliva | Baseline
  Analysis of melatonin levels by ELISA kit. Values expressed in pg/ml
Melatonin levels in plasma | Baseline
  Analysis of melatonin levels by ELISA kit. Values expressed in pg/ml
Melatonin levels in cerebrospinal fluid | Baseline
  Analysis of melatonin levels by ELISA kit. Values expressed in pg/ml

SECONDARY OUTCOMES:
Orexin levels in cerebrospinal fluid | Baseline
  Analysis of orexin levels by ELISA kit. Values expressed in ng/ml
Neurofilaments light chain levels (NFL) in cerebrospinal fluid | Baseline
  Analysis of NFL levels by SIMOA kit. Values expressed in pg/ml

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano - S. Giuseppe Hospital, Verbania, VB, Italy